CLINICAL TRIAL: NCT07285876
Title: The Effect of Sacroiliac and Lumbar Mobilizations Applied in Addition to Conventional Physical Therapy on Pain, Balance, Neuromuscular Control, and Function in Patients With Femoroacetabular Impingement Syndrome
Brief Title: The Effect of Sacroiliac and Lumbar Mobilizations Applied in Addition to Conventional Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Baha Naci, Assist Prof., Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-06/04
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Femoroacetabular Impingement Syndrome
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Group (Experimental)
  Interventions: Other: Lumbosacral Mobilization; Other: Conventional physical therapy
- Conventional Physical Therapy Group (Active Comparator)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Lumbosacral Mobilization — Sacroiliac joint: anterior ilium technique. The practitioner stabilized the sacrum. The fingers of the hand on the same side as the affected side were placed on the anterior iliac spine and the ilium was pulled upward over the sacrum.
  Sacroiliac joint: posterior ilium technique. While the patient was lying prone, the affected side was determined using the spring test. The practitioner positioned the thenar eminence of the hand against the posterior protrusion of the ilium and applied a lateral push. While maintaining this push, the patient was asked to perform backward extension.
  Lumbar region: Maitland postero-anterior technique. Grade II-III mobilization was applied to the lumbar region (L1-L5) in the postero-anterior direction. The practitioner placed the ulnar side of their hand, on the spinous process of the of the relevant segment with the wrist in extension. Using body weight, passive oscillations were performed directly on the relevant segment in the posteroanterior direction.
  Arms: Mobilization Group
Other: Conventional physical therapy — The conventional physical therapy applied to the control group included pain-targeted electrotherapy methods (Conventional transcutaneous electrical nerve stimulation, ice therapy, ultrasound therapy), hip mobilization techniques, hip strengthening exercises, core and trunk stabilization exercises, posture exercises, activity modification, and patient education.

SUMMARY:
Femoroacetabular impingement (FAI) is defined as impingement caused by abnormal morphology between the femoral head-neck junction and the acetabulum in the hip joint (Aoyama et al., 2017). As a result of morphological changes, abnormal contact between the proximal femur and acetabulum leads to chondrolabral lesions and secondary hip osteoarthritis (Casartelli, Maffiuletti, Leunig, 2019; Pierannunzii L., 2017). Femoroacetabular impingement syndrome (FAIS) is a clinical condition characterized by movement-related hip-groin pain that limits daily and athletic activities, accompanied by clinical findings, symptoms, and radiological findings associated with morphological changes (Brown-Taylor et al., 2022; Griffin et al., 2016). Symptoms typically appear suddenly and are associated with rotational and hip flexion movements that place stress on the joint (Nepple et al., 2013). The primary symptom is hip and/or groin pain related to movement or position. Typically, pain is related to activity during the acute phase, but in the chronic phase, it can occur with daily living activities or even at rest (Byrd, 2014; Nepple et al., 2013).

In patients with FAIS, reduced hip range of motion can be compensated by the pubic symphysis and sacroiliac joint (SIJ), and as a result of this compensation, hip dysfunction may develop due to increased stress on these structures. Studies describing the relationship between SIJ and FAIS are available in the literature. SIJ dysfunction causes asymmetry between the right and left innominate bones, altering the pelvic tilt angle. Excessive coverage of the femoral head by the acetabulum increases compression and creates a basis for labral tears. A study comparing postoperative pain and hip function in FAIS patients with and without SIJ anomalies showed that the group with SIJ anomalies had worse outcomes (Krishnamoorty et al., 2019).

In recent years, studies suggesting that pelvic posture and kinematics influence acetabular orientation have been increasing alongside the hip-spine concept (Krishnamoorty et al., 2019; Pierannunzii L., 2017). Although there are many similar studies in the literature examining the relationship between FAIS and the lumbopelvic junction, studies examining treatment options do not include a treatment approach targeting this relationship. While many researchers accept the value of conservative treatment methods for FAIS, there is insufficient published evidence on how this treatment should be applied.

This study was planned to investigate the effects of sacroiliac and lumbar mobilization as additional interventions to conventional physiotherapy on pain, balance, neuromuscular control, hip range of motion and hip function in patients with FAIS. The aim of our study was to include the surrounding joints that affect hip joint mechanics, as described in the literature, in the treatment program alongside physiotherapy applications, which are one of the conservative treatment methods. We also aimed to address the biomechanical limitations contributing to hip pain and dysfunction through a patient-centered approach and to evaluate their effect on the overall integrity and function of the hip and lumbopelvic joints and to evaluate its effect on the overall integrity and function of the hip and lumbopelvic joints. This study is the first to our knowledge and aims to shed light on whether patients with FAIS require more comprehensive manual therapy approaches based on the data obtained from the research.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with femoroacetabular impingement syndrome by the same orthopedic surgeon
* Having hip pain associated with femoroacetabular impingement syndrome
* Having femoroacetabular impingement syndrome morphology in the imaging methods used for femoroacetabular impingement syndrome diagnosis (Radiography, Magnetic Resonance Imaging, Computed Tomography)
* Having improved cognitive function and be willing to participate in the study
* Having signed the informed consent form

Exclusion Criteria:

* Having received physical therapy for hip pathology within the last 3 months
* Having a history of lower limb and lumbar region surgery
* Having advanced hip osteoarthritis
* Having neurological findings such as radiculopathy or myelopathy
* Having rheumatic diseases (ankylosing spondylitis, rheumatoid arthritis)
* Having infectious diseases (sacroiliitis)
* History of developmental and congenital hip dysplasia
* Fracture
* Pregnancy

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Normal Range of Hip Flexion at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  The normal range of motion of the hip joint was assessed using a universal goniometer. The patient was in the supine position while the movement was assessed. The movement being tested was demonstrated to the patient prior to measurement, and then the test was performed. When assessing hip flexion, the side being assessed was in knee flexion, while the other leg was in extension. The researcher stood beside the patient on the relevant side. The pivot point of the goniometer was placed on the patient's trochanter major. The fixed arm was placed toward the vertebral column, and the movable arm followed the lateral aspect of the femur. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Normal Range of Hip Extention at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  The normal range of motion of the hip joint was assessed using a universal goniometer. The movement being tested was demonstrated to the patient prior to measurement, and then the test was performed. When assessing hip extension, the patient was in the prone position. The pivot point of the goniometer was placed on the patient's trochanter major. The fixed arm was placed toward the vertebral column, and the movable arm followed the lateral aspect of the femur. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Normal Range of Hip Abduction at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  The normal range of motion of the hip joint was assessed using a universal goniometer. The patient was in the supine position while the hip abduction was assessed. The movement being tested was demonstrated to the patient prior to measurement, and then the test was performed. The researcher is beside the patient on the side being measured. The pivot point of the goniometer was placed on the projection of the trochanter major on the anterior surface of the femur. The fixed arm of the goniometer was held parallel to the anterior superior iliac spines. The movable arm followed the anterior midline of the femur. Attention was paid to avoid hip internal and external rotation when measuring. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Normal Range of Hip Adduction at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  The normal range of motion of the hip joint was assessed using a universal goniometer. The patient was in the supine position while the hip adduction was assessed. The movement being tested was demonstrated to the patient prior to measurement, and then the test was performed. The researcher is beside the patient on the side being measured. The pivot point of the goniometer was placed on the projection of the trochanter major on the anterior surface of the femur. The fixed arm of the goniometer was held parallel to the anterior superior iliac spines. The movable arm followed the anterior midline of the femur. Attention was paid to avoid hip internal and external rotation when measuring. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Normal Range of Hip External Rotation at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  When assessing hip external rotation, the patient is seated at the edge of the bed with knees flexed at 90°. The pivot point of the goniometer was placed on the tibial tuberosity. The fixed arm of the goniometer was positioned parallel to the floor. The movable arm followed the tibial crest. During measurement, care was taken to ensure there was no flexion, extension, abduction, or adduction movement in the hip. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Normal Range of Hip Internal Rotation at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  When assessing hip internal rotation, the patient is seated at the edge of the bed with knees flexed at 90°. The pivot point of the goniometer was placed on the tibial tuberosity. The fixed arm of the goniometer was positioned parallel to the floor. The movable arm followed the tibial crest. During measurement, care was taken to ensure there was no flexion, extension, abduction, or adduction movement in the hip. Three measurements were taken to assess joint movement. The average of the measurements was recorded.
Change from Baseline in the Pain Severity at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  The Numeric Pain Scale (NPS) was used to assess pain. The NPS is a numerical measurement tool used to subjectively assess pain intensity. The scale is numbered from 0 to 10 on a horizontal line. '0' means no pain, '5' means moderate pain, and '10' means unbearable pain. The patients were asked to assess their pain based on the pain they experienced in the last 24 hours.
Change from Baseline in the Hip Function at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  Hip function level was assessed using the Hip Outcome Score (HOS). The HOS is a 26-item measure. This scale consists of 2 separate subscales. The subscale assessing activities of daily living consists of 19 questions. Seventeen of the questions were scored and evaluated out of 68 points. The subscale assessing sports activities consists of 9 questions. All 9 questions are included in the score and evaluated out of 36 points. The HOS is measured as a percentage using the daily living activities subscale (daily living activity score/68x100) and the sports activity subscale (sports activity score/36x100) and the total HOS score (Daily Living Activity Score + Sports Activity Score/104x100) were measured as a percentage.
Change from Baseline in the Neuromuscular Control and Balance at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  Neuromuscular control and balance were assessed using a modified version of the Star Excursion Balance Test (SEBT). The SEBT used in our study was modified to include the relevant aspects of hip function. Metric measuring tapes were affixed to a flat surface so that there was a 90° angle between the posterolateral and posteromedial directions and a 135° angle between the anterior and posterior directions. The participant stood at the midpoint of the metric measuring tapes. Before starting the test, each participant was taught the test requirements with 4 trials. Participants were given a 5-minute rest period after the trials before proceeding to the test. The participant was asked to extend as far as possible in the anterior, posteromedial, and posterolateral directions with one foot on the ground and the other foot in the air, then return to the starting position. After completing 3 error-free trials in each direction, the average of these measurements was recorded in centimeters.

SECONDARY OUTCOMES:
Change from Baseline in the Lumbar and Sacroiliac Joint Mobility at 6 Weeks | From enrollment to the end of treatment at 6 weeks
  Lumbar region and sacroiliac joint mobility were assessed using the modified Schober test. While the subject stood upright, a line connecting both superior posterior iliac spines was marked 10 cm above and 5 cm below. The subject was asked to bend forward as far as possible without bending the knees. The distance between the two marked points was measured, and the difference between the measurements in the upright position and the flexion position was recorded in centimeters as the modified Schober test value.

CONTACTS AND LOCATIONS:
Overall Officials: Dilber Karagözoğlu Coşkunsu, Dr., Study Chair — Fenerbahce University
Locations (1):
- Sportomed Sports Medicine and Orthopedic Rehabilitation Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson AC, Karlsson H. The Star Excursion Balance Test: Criterion and divergent validity on patients with femoral acetabular impingement. Man Ther. 2016 Dec;26:104-109. doi: 10.1016/j.math.2016.07.015. Epub 2016 Aug 5. PMID 27525357
- [Background] Martin RL, Enseki KR, Draovitch P, Trapuzzano T, Philippon MJ. Acetabular labral tears of the hip: examination and diagnostic challenges. J Orthop Sports Phys Ther. 2006 Jul;36(7):503-15. doi: 10.2519/jospt.2006.2135. PMID 16881467
- [Background] Casartelli NC, Valenzuela PL, Maffiuletti NA, Leunig M. Effectiveness of Hip Arthroscopy on Treatment of Femoroacetabular Impingement Syndrome: A Meta-Analysis of Randomized Controlled Trials. Arthritis Care Res (Hoboken). 2021 Aug;73(8):1140-1145. doi: 10.1002/acr.24234. Epub 2021 Jul 5. PMID 32339441
- [Background] Sharma A, Alahmari K, Ahmed I. Efficacy of Manual Therapy versus Conventional Physical Therapy in Chronic Low Back Pain Due to Lumbar Spondylosis. A Pilot Study. Med Sci (Basel). 2015 Jun 26;3(3):55-63. doi: 10.3390/medsci3030055. PMID 29083391
- [Background] Ali MN, Sethi K, Noohu MM. Comparison of two mobilization techniques in management of chronic non-specific low back pain. J Bodyw Mov Ther. 2019 Oct;23(4):918-923. doi: 10.1016/j.jbmt.2019.02.020. Epub 2019 Feb 28. PMID 31733783
- [Background] Byrd JW. Femoroacetabular impingement in athletes: current concepts. Am J Sports Med. 2014 Mar;42(3):737-51. doi: 10.1177/0363546513499136. Epub 2013 Aug 27. PMID 23982400
- [Background] Krishnamoorthy VP, Beck EC, Kunze KN, Cancienne JM, Krivicich LM, Suppauksorn S, Ayeni OR, Nho SJ. Radiographic Prevalence of Sacroiliac Joint Abnormalities and Clinical Outcomes in Patients With Femoroacetabular Impingement Syndrome. Arthroscopy. 2019 Sep;35(9):2598-2605.e1. doi: 10.1016/j.arthro.2019.03.030. PMID 31500745
- [Background] Brown-Taylor L, Bordner H, Glaws K, Vasileff WK, Walrod B, Di Stasi S. Prevalence of low back pain and related disability in patients with femoroacetabular impingement syndrome. PM R. 2022 Jan;14(1):8-18. doi: 10.1002/pmrj.12572. Epub 2021 May 1. PMID 33583131
- [Background] Pierannunzii L. Pelvic posture and kinematics in femoroacetabular impingement: a systematic review. J Orthop Traumatol. 2017 Sep;18(3):187-196. doi: 10.1007/s10195-016-0439-2. Epub 2017 Feb 1. PMID 28150180
- [Background] Aoyama M, Ohnishi Y, Utsunomiya H, Kanezaki S, Takeuchi H, Watanuki M, Matsuda DK, Uchida S. A Prospective, Randomized, Controlled Trial Comparing Conservative Treatment With Trunk Stabilization Exercise to Standard Hip Muscle Exercise for Treating Femoroacetabular Impingement: A Pilot Study. Clin J Sport Med. 2019 Jul;29(4):267-275. doi: 10.1097/JSM.0000000000000516. PMID 31241527
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40989937/